CLINICAL TRIAL: NCT05691725
Title: Evaluation of Peripheral Neutrophils in Patients With Antisynthetase Syndrome
Brief Title: Evaluation of Peripheral Neutrophils in Antisynthetase Syndrome
Acronym: NEUTROSAS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI209
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Antisynthetase Syndrome
MeSH Terms: conditions — Antisynthetase syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with antisynthetase syndrome

SUMMARY:
Antisynthetase syndrome (AS) is a rare overlapping myositis characterized by cellular and humoral autoimmune responses directed against aminoacyl-tRNA synthetases. A pathogenic role of neutrophils was described during inflammatory myopathies, with increased netosis correlated with disease activity and muscle damage. Higher number of alveolar neutrophils was observed in patients with rapidly progressive forms of interstitial lung disease.

Peripheral neutrophils could represent a simple biomarker of severity and activity in patients with antisynthetase syndrome.

The main objective is to compare circulating neutrophils between severe and non severe patients with antisynthetase syndrome. Secondary objectives are: 1) to evaluate correlation between circulating neutrophils and organ-specific severity, 2) to compare circulating neutrophils at time of diagnosis and circulating neutrophils after 6 months of treatment in patients with antisynthetase syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with antisyntheatse syndrome according to Solomon criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with antisynthetase syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Number of circulating neutrophils | at diagnosis (Day 0)
  circulating neutrophils values (number of cells/mm3)
Global severity | at diagnosis (Day 0)
  composite criteria of global severity: severe interstitial lung disease (ILD) and/or severe muscular disease

SECONDARY OUTCOMES:
Circulating neutrophils change over time | at 6 months of follow-up
  circulating neutrophils values (number of cells/mm3)
ILD severity | at diagnosis (Day 0)
  %predicted FVC values in patients with ILD
ILD severity | at diagnosis (Day 0)
  %predicted DLCO values in patients with ILD
Muscular severity | at diagnosis (Day 0)
  manual muscle testing (MMT) grading in patients muscle involvement
Muscular severity | at diagnosis (Day 0)
  CPK values (U/L) in patients muscle involvement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No